CLINICAL TRIAL: NCT00024154
Title: A Phase I/II Trial of Herceptin and ZD1839 (Iressa, NSC #715055, IND#61187) in Patients With Metastatic Breast Cancer That Overexpresses HER2/Neu (erbB-2)
Brief Title: Trastuzumab and Gefitinib in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02411; E1100; U10CA021115 (NIH); CDR0000068896 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Trastuzumab; Gefitinib

ARMS (1):
- Treatment (trastuzumab, gefitinib) (Experimental): Phase I (completed): Patients receive trastuzumab (Herceptin) IV over 30-90 minutes once weekly and oral gefitinib once daily beginning on day 1.
  Cohorts of 3-6 patients receive escalating doses of gefitinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is established, additional patients are accrued to the phase II portion of the study and are treated at that dose.
  Phase II: Patients receive oral gefitinib once daily (at the MTD established in phase I) and trastuzumab IV weekly until week 24, at which time trastuzumab is given every 3 weeks (with daily gefitinib) until disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Drug: gefitinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Drug: gefitinib — Given orally
  Other Names: Iressa; ZD 1839
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving trastuzumab together with gefitinib works in treating patients with HER2-positive breast cancer. The monoclonal antibody trastuzumab can locate breast cancer cells that have HER2 on their surface and either kill them or deliver tumor-killing substances to them without harming normal cells. Biological therapies such as gefitinib may also interfere with the growth of tumor cells and may enhance the effects of trastuzumab. Combining trastuzumab with gefitinib may be an effective treatment for metastatic breast cancers with high amounts of HER2

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate, duration of response, and time to progression in patients with metastatic breast cancer that overexpresses HER2-neu treated with trastuzumab (Herceptin) and gefitinib.

II. Determine the phase II dose of gefitinib when given in combination with trastuzumab in these patients.

III. Determine the toxicity of this regimen in these patients. IV. Determine the 3- and 6-month progression-free survival of patients treated with this regimen.

V. Correlate response rates with plasma levels of circulating HER2 and tumor levels of epidermal growth factor receptor, activated HER2, and HER2 receptors, as measured by immunohistochemistry and/or fluorescent in situ hybridization (FISH), in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of gefitinib. The phase I portion of this study was open in only 5 ECOG institutions. The phase I portion has been completed, and the study is being opened in all ECOG-affiliated institutions.

Phase I (completed): Patients receive trastuzumab (Herceptin) IV over 30-90 minutes once weekly and oral gefitinib once daily beginning on day 1.

Cohorts of 3-6 patients receive escalating doses of gefitinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is established, additional patients are accrued to the phase II portion of the study and are treated at that dose.

Phase II: Patients receive oral gefitinib once daily (at the MTD established in phase I) and trastuzumab IV weekly until week 24, at which time trastuzumab is given every 3 weeks (with daily gefitinib) until disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months until 2 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic adenocarcinoma of the breast

  * Patients may have had or not had standard first-line chemotherapy for the treatment of metastatic disease
* Overexpression of HER2-neu (HER2 3+ by immunohistochemistry or gene amplification as measured by fluorescent in situ hybridization)
* Measurable disease
* Patients with no prior adjuvant chemotherapy may have failed or not failed first-line chemotherapy for metastatic disease
* No more than 2 prior systemic chemotherapy regimens for metastatic disease

  * Relapse while receiving or within 6 months of completion of adjuvant chemotherapy is considered failure of 1 regimen for metastatic disease
* No untreated brain metastases or brain metastases undergoing radiotherapy

  * Previously treated brain metastasis that has responded to radiotherapy and/or surgery allowed if not sole site of measurable disease
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - ECOG 0-2
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 3 times ULN (5 times ULN if liver metastases is present)
* INR no greater than 1.5 times ULN
* PT and PTT no greater than 1.5 times ULN
* Creatinine no greater than 1.5 mg/dL
* No more than trace blood or protein in urine
* LVEF ≥ 50% by MUGA scan
* No prior New York Heart Association class I-IV heart disease
* No PR prolongation or atrioventricular block on ECG
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception (preferably nonhormonal)
* Random blood sugar less than 2.5 times ULN
* No other malignancy within the past 5 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other acute or chronic medical or psychiatric condition or laboratory abnormality that would preclude study participation
* No prior trastuzumab (Herceptin)
* No other concurrent immunologic therapy
* See Disease Characteristics
* Recovered from prior cytotoxic chemotherapy
* No prior cumulative dose of doxorubicin more than 360 mg/m^2
* No concurrent chemotherapy
* At least 2 weeks since prior hormonal therapy
* No concurrent hormonal therapy, including tamoxifen
* No concurrent dexamethasone, progesterone, or glucocorticoids
* See Disease Characteristics
* At least 2 weeks since prior radiotherapy
* No prior radiotherapy to target lesions or only site of measurable disease
* No concurrent radiotherapy
* See Disease Characteristics
* No prior organ allograft
* No prior gefitinib
* No prior immunosuppressive therapy
* At least 2 weeks since prior cytotoxic drugs
* No concurrent carbamazepine, ethosuximide, griseofulvin, nafcillin, nelfinavir mesylate, nevirapine, oxcarbazepine, phenobarbital, phenylbutazone, phenytoin, primidone, rifabutin, rifampin, rofecoxib, Hypericum perforatum (St. John's Wort), sulfadimidine, sulfinpyrazone, troglitazone, or grapefruit juice
* No other concurrent investigational agents
* No concurrent topical eye agents
* Concurrent bisphosphonates allowed for hypercalcemia and/or prophylaxis of bone metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2002-02; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
MTD and DLT in patients treated with Herceptin and ZD1839 graded using the NCI CTC (Phase I) | 4 weeks

SECONDARY OUTCOMES:
Median time to progression (Phase II) | 6 months
Progression-free survival (Phase II) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Arteaga, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States